CLINICAL TRIAL: NCT06424509
Title: Effects of Psychiatric Admissions on Self-harm and Suicide in People With Borderline Personality Disorder
Status: Recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-00589-01
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Borderline Personality Disorder; Self-harm; Non-suicidal Self-injury; Suicide
MeSH Terms: conditions — Borderline Personality Disorder; Self-Injurious Behavior; Suicide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High admission: The quartile of participants using the highest degree of long (>5 days) and/or compulsory psychiatric inpatient care.
  Interventions: Other: High degree of long (>5 days) and/or compulsory psychiatric inpatient care
- Low admission: The quartile of participants using the lowest degree of long (>5 days) and/or compulsory psychiatric inpatient care.

INTERVENTIONS:
Other: High degree of long (>5 days) and/or compulsory psychiatric inpatient care — High degree of long (>5 days) and/or compulsory psychiatric inpatient care
  Groups: High admission

SUMMARY:
The current study aims to evaluate the impact of long (>5 days) and/or compulsory psychiatric inpatient care on subsequent healthcare utilization for self-harm and suicide in people with borderline personality disorder, a condition characterized by frequent self-harm.

The basis for this study is the diversity of clinical practices across Swedish regions. By categorizing clinics based on their practices with respect to long and/or compulsory psychiatric inpatient care, it is possible to explore the impact of these practices on subsequent somatic and psychiatric healthcare, including emergency care due to self-harm as well as on completed suicides.

All psychiatric clinics across Sweden authorized to administer compulsory care for adults, totalling 78 clinics will be included. Each clinic per specific calendar year will represent one participant, identified by the clinic's name and the respective year (e.g., Umeå2010, Linköping2013, Malmö2022).

Data collection will involve the utilization of the national registers to capture outcome measures and account for confounding factors. The participants will be ranked based on a composite variable, which includes the average number of days spent in inpatient compulsory care and other psychiatric inpatient care exceeding 5 days, among individuals diagnosed with BPD. The top quartile of participants will be compared with the bottom quartile.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric clinic in Sweden authorized to administer compulsory care for adults. Each clinic per specific calendar year will represent one participant, identified by the clinic's name and the respective year (e.g., Umeå2010, Linköping2013, Malmö2022).

Exclusion Criteria:

* No authorization to administer compulsory care for adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All psychiatric clinics across Sweden authorized to administer compulsory care for adults, totalling 78 clinics. Each clinic per specific calendar year will represent one participant, identified by the clinic's name and the respective year (e.g., Umeå2010, Linköping2013, Malmö2022).
Sampling Method: Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of healthcare visits due to self-harm | 1 year
  Number of healthcare visits due to self-harm in specialized inpatient or outpatient care, as defined in the NPR (X60-X84; Intentional self-harm) divided by the number of individuals diagnosed with BPD per clinic and calendar year.
Number of deaths by suicide | 1 year
  Number of deaths by suicide (X60-X84; Intentional self-harm or Y10-34; Events of undetermined intent) in individuals diagnosed with BPD divided by the number of individuals diagnosed with BPD per clinic and calendar year.
Number of deaths by suicide within 30 days after discharge | 1 year
  Number of deaths by suicide (X60-X84; Intentional self-harm or Y10-34; Events of undetermined intent) within 30 days after discharge, in individuals diagnosed with BPD divided by the number of individuals diagnosed with BPD, per clinic and calendar year

SECONDARY OUTCOMES:
Number of days between admissions to psychiatric inpatient care | 1 year
  Number of days between admissions to psychiatric inpatient care for people diagnosed with BPD divided by the number of individuals diagnosed with BPD per clinic and calendar year.
Number of days between death by suicide and discharge | 1 year
  Number of days between death by suicide (X60-X84; Intentional self-harm or Y10-34; Events of undetermined intent) and discharge in individuals diagnosed with BPD. For this variable, death by suicide during inpatient admission will be labelled 0.
Number of days in somatic (non-psychiatric) inpatient care after self-harm | 1 year
  Number of days in somatic (non-psychiatric) inpatient care after self-harm (X60-X84; Intentional self-harm) divided by the number of individuals diagnosed with BPD per clinic and calendar year.

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Westling, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Sweden

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT06424509/Prot_SAP_000.pdf